CLINICAL TRIAL: NCT01678846
Title: The Good Schools Study: Cluster Randomised Controlled Trial of a Program to Prevent Violence Against Children in Schools
Brief Title: Good Schools Study
Acronym: GSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Raising Voices (Other); Institute of Education, UK (Unknown); Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LSHTM_6183
Record Dates: First submitted 2012-08-24; First posted 2012-09-05 (Estimated); Results first posted 2016-01-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2015-06

CONDITIONS: Physical Violence; Educational Achievement; Mental Health; Sexual Violence; Violence Against Children
Keywords: corporal punishment; violence; education; depression; anxiety; conduct disorder
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders; Conduct Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Good School Toolkit (Experimental): Schools in the intervention arm will receive the Good Schools Toolkit materials and implementation support.
  Interventions: Behavioral: Good School Toolkit
- Control (No Intervention): Schools in this arm will receive the Good Schools Toolkit materials and some implementation support after the end of the trial.

INTERVENTIONS:
Behavioral: Good School Toolkit — The Toolkit uses a six step process to create a school wide intervention that engages teachers, students, administration, and parents to reflect on how they can promote quality of education in their school. The Toolkit articulates complex ideas (what is a good learning environment, a good teacher, how to create positive discipline without using violence) through booklets, posters and school initiated learning processes. Specific modules on alternative discipline techniques and how staff can use positive discipline are included in the Toolkit. The intervention includes sessions on knowledge, attitudes and opportunities to practice new behavioural skills. Work is led by teachers and students, and supported by visits from Raising Voices staff. The Toolkit can be reviewed at (http://www.raisingvoices.org/children/good_school_toolkit.php).
  Arms: Good School Toolkit

SUMMARY:
The purpose of this study is to determine whether use of the Good Schools Toolkit is effective in reducing violence against children in primary schools.

DETAILED DESCRIPTION:
Violence against children has profound effects on both children's health and their ability to do well at school. Fear, anxiety and injuries caused by violence may play a large role in both children's absenteeism and low educational achievement, and there is increasing interest from large bilateral donors in investigating this link in low income countries. The Good School Toolkit has been developed and refined for 6 years in Uganda by Raising Voices. The toolkit takes a systemic approach, involving an entire school in a process of change to reduce violence and improve teaching techniques. The Toolkit draws on the Transtheoretical Model and incorporates standard behaviour change techniques such as setting a goal and making an action plan, which are effective in modifying behaviour. This study aims to determine whether use of the Good School Toolkit reduces children's experience of violence by school staff. The investigators will also examine the effects of the Toolkit on children's educational outcomes, mental health and well-being.

The investigators will conduct a cluster randomised controlled trial in 40 primary schools in Luwero District, Uganda. More than 3500 children in Primary 5, 6 and 7 will be surveyed (aged about 11-16 years). Half of the schools will receive the Toolkit, and other half will be put on a waiting list to receive the Toolkit at the end of the study. The results from this evaluation will be used to brief policy-makers within the Ministry of Education and Sports involved in developing country-wide policy and practice around violence against children in schools.

ELIGIBILITY:
1. Inclusion Criteria:

   * Schools

     * in Luwero District, Uganda
     * more than 40 students registered in Primary 5
   * Participants

     * registered as a Primary 5, 6 or 7 pupil
     * any school staff member
2. Exclusion Criteria:

   * Schools

     -- existing program related to prevention of violence against children or school governance
   * Participants -- not able to understand consent and study procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3820 (Actual)
Dates: Start 2012-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Devries, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- District-wide, Multiple, Luwero District, Uganda

REFERENCES:
- [Derived] Knight L, Atuhaire L, Bhatia A, Allen E, Namy S, Anton-Erxleben K, Nakuti J, Mirembe A, Nakiboneka M, Seeley J, Weiss HA, Parkes J, Bonell C, Naker D, Devries K. Violence outcomes in later adolescence with the Good School Toolkit-Primary: a nonrandomized controlled trial in Uganda. BMC Public Health. 2024 Jun 7;24(1):1532. doi: 10.1186/s12889-024-19024-5. PMID 38849782
- [Derived] Carlson C, Namy S, Norcini Pala A, Wainberg ML, Michau L, Nakuti J, Knight L, Allen E, Ikenberg C, Naker D, Devries K. Violence against children and intimate partner violence against women: overlap and common contributing factors among caregiver-adolescent dyads. BMC Public Health. 2020 Jan 29;20(1):124. doi: 10.1186/s12889-019-8115-0. PMID 31996179
- [Derived] Devries K, Parkes J, Knight L, Allen E, Namy S, Datzberger S, Nalukenge W, Atuhaire L, Kyegombe N, Walakira E, Seeley J, Weiss HA, Naker D. Context of Violence in Adolescence Cohort (CoVAC) study: protocol for a mixed methods longitudinal study in Uganda. BMC Public Health. 2020 Jan 13;20(1):43. doi: 10.1186/s12889-019-7654-8. PMID 31931768
- [Derived] Knight L, Allen E, Mirembe A, Nakuti J, Namy S, Child JC, Sturgess J, Kyegombe N, Walakira EJ, Elbourne D, Naker D, Devries KM. Implementation of the Good School Toolkit in Uganda: a quantitative process evaluation of a successful violence prevention program. BMC Public Health. 2018 May 9;18(1):608. doi: 10.1186/s12889-018-5462-1. PMID 29743105
- [Derived] Devries K, Kuper H, Knight L, Allen E, Kyegombe N, Banks LM, Kelly S, Naker D. Reducing Physical Violence Toward Primary School Students With Disabilities. J Adolesc Health. 2018 Mar;62(3):303-310. doi: 10.1016/j.jadohealth.2017.09.004. Epub 2017 Dec 6. PMID 29217214
- [Derived] Kayiwa J, Clarke K, Knight L, Allen E, Walakira E, Namy S, Merrill KG, Naker D, Devries K. Effect of the good school toolkit on school staff mental health, sense of job satisfaction and perceptions of school climate: Secondary analysis of a cluster randomised trial. Prev Med. 2017 Aug;101:84-90. doi: 10.1016/j.ypmed.2017.05.022. Epub 2017 Jun 2. PMID 28579503
- [Derived] Grundlingh H, Knight L, Naker D, Devries K. Secondary distress in violence researchers: a randomised trial of the effectiveness of group debriefings. BMC Psychiatry. 2017 Jun 2;17(1):204. doi: 10.1186/s12888-017-1327-x. PMID 28578682
- [Derived] Devries KM, Knight L, Child JC, Kyegombe N, Hossain M, Lees S, Watts C, Naker D. Witnessing intimate partner violence and child maltreatment in Ugandan children: a cross-sectional survey. BMJ Open. 2017 Feb 28;7(2):e013583. doi: 10.1136/bmjopen-2016-013583. PMID 28246136
- [Derived] Thumann BF, Nur U, Naker D, Devries KM. Primary school students' mental health in Uganda and its association with school violence, connectedness, and school characteristics: a cross-sectional study. BMC Public Health. 2016 Jul 29;16:662. doi: 10.1186/s12889-016-3351-z. PMID 27473040
- [Derived] Clarke K, Patalay P, Allen E, Knight L, Naker D, Devries K. Patterns and predictors of violence against children in Uganda: a latent class analysis. BMJ Open. 2016 May 24;6(5):e010443. doi: 10.1136/bmjopen-2015-010443. PMID 27221125
- [Derived] Devries KM, Child JC, Elbourne D, Naker D, Heise L. "I never expected that it would happen, coming to ask me such questions":Ethical aspects of asking children about violence in resource poor settings. Trials. 2015 Nov 11;16:516. doi: 10.1186/s13063-015-1004-7. PMID 26558829
- [Derived] Devries KM, Knight L, Child JC, Mirembe A, Nakuti J, Jones R, Sturgess J, Allen E, Kyegombe N, Parkes J, Walakira E, Elbourne D, Watts C, Naker D. The Good School Toolkit for reducing physical violence from school staff to primary school students: a cluster-randomised controlled trial in Uganda. Lancet Glob Health. 2015 Jul;3(7):e378-86. doi: 10.1016/S2214-109X(15)00060-1. PMID 26087985
- [Derived] Child JC, Naker D, Horton J, Walakira EJ, Devries KM. Responding to abuse: Children's experiences of child protection in a central district, Uganda. Child Abuse Negl. 2014 Oct;38(10):1647-58. doi: 10.1016/j.chiabu.2014.06.009. Epub 2014 Jul 14. PMID 25035172
- [Derived] Devries KM, Allen E, Child JC, Walakira E, Parkes J, Elbourne D, Watts C, Naker D. The Good Schools Toolkit to prevent violence against children in Ugandan primary schools: study protocol for a cluster randomised controlled trial. Trials. 2013 Jul 24;14:232. doi: 10.1186/1745-6215-14-232. PMID 23883138

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cross-sectional baseline and endline surveys were conducted in 42 schools in June/July 2012 and June/July 2014. A simple random sample of up to 130 P5, 6 and 7 students were invited for individual interviews. If there were fewer than 130 P5-7 students in a school, all were invited for interview.
Period: Overall Study
Arm/Group | Good School Toolkit | Control
Started | 1921 (Whole school implementation. Started and completed shows number of students in the end-line survey.) | 1899
Completed | 1921 | 1899
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline survey total participants is shown here (whereas the number in the participant flow is the number of participants at endline, in both the "started and "completed")
Groups:
- Total: Total of all reporting groups
Arm/Group | Good School Toolkit | Control | Total
Number analyzed (Participants) | 1824 | 1882 | 3706
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.1 (1.5) | 13.0 (1.5) | 13.0 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 927 | 1010 | 1937
  Male | 897 | 872 | 1769

OUTCOME MEASURES:

1. Primary Outcome: Physical Violence From School Staff
Description: past week experience of any physical violence from school staff
Time Frame: 2-year follow-up
Measure: Number; unit: participants
Arm/Group | Good School Toolkit | Control
Number analyzed (Participants) | 1921 | 1899
participants | 595 | 924
Statistical Analysis 1: Comparison: Good School Toolkit vs Control; Does the Toolkit intervention reduce physical violence from school staff to Ugandan primary school students; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.26 to 0.64] — An odds ratio of less than 1 would demonstrate a protective effect of the intervention. Unadjusted odds ratio presented, accounting for correlation between students within schools

2. Secondary Outcome: Child Mental Health
Description: score on the Strengths and Difficulties Questionnaire (SDQ): 20 questions. Total difficulties score, divided by the number of completed items. Modelled as a continuous variable. Range 0 (no difficulties) to 2 (high difficulties).
Time Frame: 2-year follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Good School Toolkit | Control
Number analyzed (Participants) | 1921 | 1899
units on a scale | 0.44 (0.26) | 0.44 (0.26)

3. Secondary Outcome: Educational Achievement: Word Recognition in English
Description: Word recognition in English(words per minute). Early Grade Reading Assessment, Uganda version. Calculated as number of words read correctly (out of a maximum of 50), divided by the time (out of a maximum of 60 seconds).
Time Frame: 2-year follow-up
Measure: Mean (Standard Deviation); unit: words per minute
Arm/Group | Good School Toolkit | Control
Number analyzed (Participants) | 1921 | 1899
words per minute | 48.6 (27.7) | 49.7 (27.7)

4. Secondary Outcome: Safety and Well-being at School
Description: Five questions. Each question asked with response options: all the time, most of the time, sometimes, never:
  I feel that my teachers care about me. I feel safe in school. I feel like I belong at school. I like to spend time at school. I am scared of my teachers (reverse coded). Scores summed, modelled as a continuous variable. Range 0 (low) to 15 (high). Higher score is better safety and well-being at school.
Time Frame: At 2 year follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Good School Toolkit | Control
Number analyzed (Participants) | 1921 | 1899
units on a scale | 11.7 (2.4) | 11.1 (2.5)

ADVERSE EVENTS:
Arm/Group | Good School Toolkit | Control
Serious Adverse Events (participants affected / at risk) | 0/1921 | 0/1899
Other Adverse Events (participants affected / at risk) | 0/1921 | 0/1899

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes